CLINICAL TRIAL: NCT06887530
Title: Validity and Reliability of the Hand-10 Questionnaire in Children With Unilateral Cerebral Palsy
Brief Title: Hand-10 Questionnaire in Children With Unilateral Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: Hand-10 Questionnaire
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy (CP); Hand Functions
Keywords: cerebral palsy; hand functions; Questionnaire validation; Disability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Unilateral Cerebral Palsy: Children between the ages of 6-15, diagnosed with unilateral cerebral palsy, with sufficient cognitive status to understand the evaluation commands and with reading skills will be included.
  Interventions: Other: Hand-10 questionnaire and ABILHAND-kids questionnaire

INTERVENTIONS:
Other: Hand-10 questionnaire and ABILHAND-kids questionnaire — Children and their parents included in the study will be informed about the purpose of the study and the evaluations to be made and will be asked to sign a written consent form. The questions in the data collection form will be asked to individuals in a face-to-face interview. The manual skills classification system, Hand-10 questionnaire and ABILHAND-kids questionnaire will be used.
  While validating the Hand10 questionnaire in children with cerebral palsy, it was planned to use the ABILHAND-kids scale, which has been previously validated for reliability and validity in cerebral palsy. It was also planned to use the hand function classification system in the evaluations. The Hand-10 questionnaire will be filled out by the child himself. The ABILHAND-kids questionnaire will be filled out by the parent. An expert will record the manuel ability system according to the hand skills.

SUMMARY:
A Turkish version of the Hand-10 (unabbreviated) questionnaire has been developed, but its validity and reliability in cerebral palsy has not yet been proven. In particular, questioning daily life activities with visual content can make a significant contribution to evaluating hand functions and independence. Therefore, the aim of this planned study was to investigate the validity and reliability of the Hand-10 questionnaire in cerebral palsy.

DETAILED DESCRIPTION:
The Hand-10 questionnaire was developed to evaluate upper extremity problems. It is a clear, short, and visual questionnaire that the individual fills out on their own. It includes shoulder, elbow, wrist, and hand functions. The developers of the questionnaire stated that it can be easily applied to children due to its visual explanations. Pictorial materials make the survey more understandable for the elderly and children. Visual content makes participation more enjoyable, especially for children. Due to its visual content, Hand10 has been proven to be applicable to the elderly and children. For its high accuracy, it is recommended to analyze its validity in specific diseases in previous studies. However, there are only two studies to date that have shown its validity for patients with lateral epicondylitis and trigger finger. Due to its clarity and visuals, it can make a significant contribution to the assessment methods used especially in children with cerebral palsy. Therefore, investigating its validity and reliability in children with cerebral palsy can provide support to the literature and professionals working in this field.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6-15, diagnosed with unilateral cerebral palsy,
* With sufficient cognitive status to understand assessment instructions
* With reading skills

Exclusion Criteria:

* Those with health problems not related to cerebral palsy,
* neglect of the affected extremity,
* serious visual problems,
* undergoing botox or orthopedic surgery in the last 6 months,
* not willing to participate in the study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 6 and 15 who have been diagnosed with unilateral cerebral palsy and who have sufficient cognitive status to understand assessment instructions and reading skills will be included.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Manual Ability Classification System | 1-3 months
  The Manual Ability Classification System is a classification system that evaluates the hand-use skills of children with Cerebral palsy between the ages of 4 and 18 in their daily activities. It evaluates how the child holds objects on his/her own and the extent to which he/she needs assistance and adaptation when performing various functions using his/her hand in his/her daily life. It measures the general capacity to hold objects. It focuses on how the child holds objects appropriate for his/her age, regardless of the difference in function between the two hands. While Level I is the best in terms of manual skills, Level V represents the least adequate situation.
Hand-10 questionnaire | 1-3 months
  The Hand-10 (unabbreviated) questionnaire consists of 10 items. It was developed to evaluate upper extremity problems. It is a clear, short questionnaire with visual elements. It includes shoulder, elbow, wrist and hand functions. Hand-10 questionnaire assesses complaints related to hand disorders with 10 items. Patients rate their performance over the past week on a scale from 0 to 10 (0: no limitation, 10: impossible), with total scores ranging from 0 to 100. Higher scores indicate worse functional status.The presence of visual explanations allows easy application for children and the elderly. The Hand-10 questionnaire has been used to evaluate the results of lateral epicondylitis treatment and cases with carpal tunnel syndrome.
ABILHAND-kids questionnaire | 1-3 months
  ABILHAND-Kids questionnaire is a valid and reliable questionnaire developed to assess the perceived manual skills of children with cerebral palsy or their parents. It is used in children aged 6-15. The questionnaire assesses a person's daily life activities that require upper extremity function. It consists of 21 items. Each item is evaluated between 0 and 2 points (0: impossible, 1: difficult, 2: easy). A higher score indicates better upper extremity function. There is a Turkish version of the ABILHAND-kids questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurimoto S, Suzuki M, Yamamoto M, Okui N, Imaeda T, Hirata H. Development and validation of a ten-item questionnaire with explanatory illustrations to assess upper extremity disorders: favorable effect of illustrations in the item reduction process. J Orthop Sci. 2011 Nov;16(6):737-44. doi: 10.1007/s00776-011-0148-x. Epub 2011 Sep 10. PMID 21912917
- [Background] Oksuz C, Alemdaroglu I, Kilinc M, Abaoglu H, Demirci C, Karahan S, Yilmaz O, Yildirim SA. Reliability and validity of the Turkish version of ABILHAND-Kids' questionnaire in a group of patients with neuromuscular disorders. Physiother Theory Pract. 2017 Oct;33(10):780-787. doi: 10.1080/09593985.2017.1346026. Epub 2017 Jul 17. PMID 28715270
- [Background] de Jong LD, van Meeteren A, Emmelot CH, Land NE, Dijkstra PU. Reliability and sources of variation of the ABILHAND-Kids questionnaire in children with cerebral palsy. Disabil Rehabil. 2018 Mar;40(6):684-689. doi: 10.1080/09638288.2016.1272139. Epub 2017 Jan 9. PMID 28068864
- [Background] Moritomo H, Imaeda T, Gotani H, Momose T, Abe Y, Oi H, Omokawa S, Sawaizumi T, Nemoto K; Functional Evaluation Committee of Japanese Society for Surgery of Hand. Reliability of the Hand20 questionnaire: comparison with the 36-Item Short-Form Health Survey. Hand Surg. 2014;19(1):1-6. doi: 10.1142/S0218810414500014. PMID 24641733
- [Background] Kurimoto S, Yamamoto M, Shinohara T, Tatebe M, Katsuyuki I, Hirata H. Favorable effects of explanatory illustrations attached to a self-administered questionnaire for upper extremity disorders. Qual Life Res. 2013 Jun;22(5):1145-9. doi: 10.1007/s11136-012-0233-4. Epub 2012 Jul 22. PMID 22820834
- [Background] Anttila H, Autti-Ramo I, Suoranta J, Makela M, Malmivaara A. Effectiveness of physical therapy interventions for children with cerebral palsy: a systematic review. BMC Pediatr. 2008 Apr 24;8:14. doi: 10.1186/1471-2431-8-14. PMID 18435840
- [Background] Alhusaini AA, Fallatah S, Melam GR, Buragadda S. Efficacy of transcutaneous electrical nerve stimulation combined with therapeutic exercise on hand function in children with hemiplegic cerebral palsy. Somatosens Mot Res. 2019 Mar;36(1):49-55. doi: 10.1080/08990220.2019.1584555. Epub 2019 Mar 26. PMID 30913943